CLINICAL TRIAL: NCT01435317
Title: Prospective Clinical Study for Confirmation of Efficacy and Safety of Acoustic CR®-Neuromodulation by CE Marked ANM T30 CR®-System in a "Real Life" Patient Population With Chronic Tonal Tinnitus
Brief Title: Acoustic Coordinated Reset (CR®) Neuromodulation for the Treatment of Chronic Tonal Tinnitus ("RESET Real Life")
Acronym: RRL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ANM Adaptive Neuromodulation GmbH (Industry)
Collaborators: CERES GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCT2011-08-26
Record Dates: First submitted 2011-08-31; First posted 2011-09-16 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Tinnitus
Keywords: Acoustic CR®-neuromodulation; ANM T30 CR®-System
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- standard (Experimental): Standard treatment with the ANM T30 CR®-System
  Interventions: Device: ANM T30 CR®-System

INTERVENTIONS:
Device: ANM T30 CR®-System — Stimulation for 4-6h/day for a time of 1 year

SUMMARY:
Confirmation of efficacy and safety of acoustic CR®-neuromodulation for the treatment of chronic tinnitus patients using the CE marked ANM T30 CR®-system in a real life outpatient setting.

* Identification of early indicators for therapy success
* Comparison of different patient groups regarding: tinnitus severity, tinnitus duration, level of hearing loss, stimulation patterns, unilateral monotonal vs. all other complex forms
* Representative set of safety data in a broad patient spectrum
* Measurement of tinnitus burden (TBF-12 Questionnaire)
* Generation of longterm compliance data

ELIGIBILITY:
Main Inclusion Criteria:

* symptomatic subjective tonal chronical (> 3 months) tinnitus
* <60dB hearing loss
* men and women ≥18 years old

Main Exclusion Criteria:

* serious neurologic
* psychiatric or internistic disease
* objective tinnitus
* Morbus Menière
* craniomandibular triggered tinnitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Improvement of TBF-12 Score or CGI Score | 12 months
  Change of tinnitus severity, measured by TBF-12 Score or CGI score change from baseline to end of treatment.

SECONDARY OUTCOMES:
NRS loudness and annoyance (0-100) | 0.5, 1, 2, 3, 6, 9, 12 months
Tinnitus-freedom | 3,6,9,12 months
Compliance | 0.5,1,3,6,9,12 months
  Questioning if the specified application was kept.
Alteration of tinnitus | 0.5,1,2,3,6,9,12 months
  Early alteration of tinnitus frequency and psychometric tinnitus loudness, measured with the ANM T30 CR®-System.
Audiogram for hearing loss change | 3,12 months
TBF-12 | 3,6,9,12 months

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Brinkmann, Dr. med., Principal Investigator — HNO-Gemeinschaftspraxis Hamm-Ahlen-Oelde
Locations (23):
- Germany (23):
  - Dr. med. Mueller, Augsburg
  - Dr. med. Jan Loehler, Bad Bramstedt
  - Praxisverbund Berlin, Berlin
  - Dr. med. Daniel Osterland, Berlin
  - Dres. med. Bodlien/Lingner/Kassuhn, Braunschweig
  - Praxis HNO Koeln Nord, Cologne
  - Dres. Lindenberger Wilhelm Ecke Elies Sperl Brackmann, Frankfurt
  - Dr. med. Fleissner, Freiburg im Breisgau
  - EuromedClinic, Fürth
  - Dr. med. Hegemann-Gaertner, Grevenbroich
  - Dipl.-Med. Kathrin Stoelzer, Halle
  - Dr. med. Hahbrock, Koblenz
  - Dr. med. Wichmann, Krefeld
  - Roemerwallklini Gmbh, Mainz
  - HNO-Gemeinschaftspraxis im Zentrum, Mannheim
  - Dr .med. Tatjana von Stackelberg, Meerbusch
  - Dr. med. Ullmann, Melsungen
  - Dr. med. Wurzer, München
  - Dres. med. Bergmann und Davies, Nürtingen
  - Dr. med Uwe Brinkmann, Oelde
  - Dr. med. Huegelschaeffer, Philippsburg
  - Dr. med. Axel Roesler, Radevormwald
  - Dres. med. Ramming und Waller, Schweinfurt